CLINICAL TRIAL: NCT05001490
Title: Effectiveness of Smartphone Application Based Brushing Reminder Therapy for Plaque Control in Orthodontic Patients: A Randomized Controlled Trial
Brief Title: Smartphone Application Based Reminder Therapy in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, Salman Khan, Resident, department of orthodontics, Rehman Medical Institute - RMI
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EC 2020-09-055
Record Dates: First submitted 2021-04-01; First posted 2021-08-12 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Orthodontic Appliance Complication
Keywords: oral hygiene; smartphone application; plaque index

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Other: Smartphone application based reminder
- Control group (No Intervention)

INTERVENTIONS:
Other: Smartphone application based reminder — Brushing reminders were given to the patients in experimental group through a smartphone application twice daily
  Other Names: Routine oral hygiene instructions
  Arms: Experimental group

SUMMARY:
This randomized control trial was performed to asses the efficiency of smartphone application based reminder therapy on plaque control and oral hygiene at two points in time.

DETAILED DESCRIPTION:
This randomized controlled trial was performed to assess the effect of the smartphone application based reminders for oral hygiene reinforcement on orthodontic patients. Methods: 60 orthodontic patients were randomly allocated to either control or experimental group (30 each). Experimental groups received reminders twice a day by a smartphone application. Plaque scoring was done by using Turesky modified Quigley-Hein plaque index (TMQHPI) at baseline(T0), after 2 weeks(T1) and after 6 weeks(T3). Results: Significant difference in plaque scores was found at T2(6 weeks), but no significant difference was found at T1(2 weeks). Conclusions: Active smartphone-based reminder therapy for oral hygiene maintenance during fixed appliance orthodontic treatment decreases the plaque scores in patients in medium to long term

ELIGIBILITY:
Inclusion Criteria:

- A total of Sixty (60) patients between 12-30 years of age undergoing fixed appliance therapy were included in the study. All the participants had to be in at least 4 weeks of active orthodontic therapy with fixed appliances in all the quadrants of the oral cavity. Further inclusion criteria were familiarity with smartphone and a personal smartphone with Android version ≥ 6.0 or iOS version ≥ 10 operating system, good general and dental health (no active caries, no advanced gingivitis, or periodontitis needing periodontal therapy), with no history of smoking or any other form of tobacco use, no antibiotic or chlorhexidine containing mouth rinses used within two weeks of screening.

Exclusion Criteria:

- Patients with prosthesis in the mouth and those taking antibiotics, anti-epileptics, anti-hypertensives and immunosuppressive medications were excluded from the study.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Plaque index score | 0 weeks ( at T0)
  Turesky modified Quigley-Hein plaque index (score: minimum=0 maximum=5. worsening with increase in score from 0-5)
Plaque index score | 2 weeks ( at T1)
  Turesky modified Quigley-Hein plaque index (score: minimum=0 maximum=5. worsening with increase in score from 0-5)
Plaque index score | 6 weeks (at T2)
  Turesky modified Quigley-Hein plaque index (score: minimum=0 maximum=5. worsening with increase in score from 0-5)

CONTACTS AND LOCATIONS:
Overall Officials: Aneela Nausheen, FCPS, Study Chair — Rehman-MI; Muhammad K Asif, PHD, Study Chair — Rehman-MI
Locations (1):
- Rehman medical institute, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zachrisson BU. Gingival condition associated with orthodontic treatment. II. Histologic findings. Angle Orthod. 1972 Oct;42(4):353-7. No abstract available. PMID 4507151
- [Background] Parizi MT, Mohammadi TM, Afshar SK, Hajizamani A, Tayebi M. Efficacy of an electric toothbrush on plaque control compared to two manual toothbrushes. Int Dent J. 2011 Jun;61(3):131-5. doi: 10.1111/j.1875-595X.2011.00029.x. PMID 21692783
- [Background] Eppright M, Shroff B, Best AM, Barcoma E, Lindauer SJ. Influence of active reminders on oral hygiene compliance in orthodontic patients. Angle Orthod. 2014 Mar;84(2):208-13. doi: 10.2319/062813-481.1. Epub 2013 Sep 12. PMID 24028316
- [Background] Al-Jewair TS, Suri S, Tompson BD. Predictors of adolescent compliance with oral hygiene instructions during two-arch multibracket fixed orthodontic treatment. Angle Orthod. 2011 May;81(3):525-31. doi: 10.2319/092010-547.1. Epub 2011 Feb 9. PMID 21306222
- [Background] Cozzani M, Ragazzini G, Delucchi A, Mutinelli S, Barreca C, Rinchuse DJ, Servetto R, Piras V. Oral hygiene compliance in orthodontic patients: a randomized controlled study on the effects of a post-treatment communication. Prog Orthod. 2016 Dec;17(1):41. doi: 10.1186/s40510-016-0154-9. Epub 2016 Dec 19. PMID 27891568
- [Background] Erbe C, Klees V, Ferrari-Peron P, Ccahuana-Vasquez RA, Timm H, Grender J, Cunningham P, Adam R, Farrell S, Wehrbein H. A comparative assessment of plaque removal and toothbrushing compliance between a manual and an interactive power toothbrush among adolescents: a single-center, single-blind randomized controlled trial. BMC Oral Health. 2018 Aug 3;18(1):130. doi: 10.1186/s12903-018-0588-1. PMID 30075780
- [Result] Cardoso Mde A, Saraiva PP, Maltagliati LA, Rhoden FK, Costa CC, Normando D, Capelozza Filho L. Alterations in plaque accumulation and gingival inflammation promoted by treatment with self-ligating and conventional orthodontic brackets. Dental Press J Orthod. 2015 Mar-Apr;20(2):35-41. doi: 10.1590/2176-9451.20.2.035-041.oar. PMID 25992985
- [Result] McCarney R, Warner J, Iliffe S, van Haselen R, Griffin M, Fisher P. The Hawthorne Effect: a randomised, controlled trial. BMC Med Res Methodol. 2007 Jul 3;7:30. doi: 10.1186/1471-2288-7-30. PMID 17608932
- [Result] Schwebel FJ, Larimer ME. Using text message reminders in health care services: A narrative literature review. Internet Interv. 2018 Jun 21;13:82-104. doi: 10.1016/j.invent.2018.06.002. eCollection 2018 Sep. PMID 30206523
- [Result] Farhadifard H, Soheilifar S, Farhadian M, Kokabi H, Bakhshaei A. Orthodontic patients' oral hygiene compliance by utilizing a smartphone application (Brush DJ): a randomized clinical trial. BDJ Open. 2020 Nov 20;6(1):24. doi: 10.1038/s41405-020-00050-5. PMID 33298841